CLINICAL TRIAL: NCT03188003
Title: Comparison of Lumbo-pelvic Mobilization and Stabilization Exercises With Pilates Method in Non-specific Chronic Low Back Pain and Movement Functionality
Brief Title: Lumbo-pelvic Mobilization and Stabilization With Pilates Method in Low Back Pain and Movement Functionality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jefferson Fagundes Loss, Doctor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOB X STAB in Pilates
Record Dates: First submitted 2017-05-18; First posted 2017-06-15 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Low Back Pain; Pain
Keywords: Exercise Movement Techniques; Low Back Pain; Exercise
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization (Experimental): This group will undergo 10 Pilates sessions with a focus on lumbo-pelvic stabilization exercises approach.
  Intervention administered: Exercise Movement Techniques (Pilates Exercise) based on stabilization
  Interventions: Other: Exercise Movement Techniques based on stabilization
- Mobilization (Experimental): This group will undergo 10 Pilates sessions with a focus on lumbo-pelvic mobilization exercises approach.
  Intervention administered: Exercise Movement Techniques (Pilates Exercise) based on mobilization
  Interventions: Other: Exercise Movement Techniques based on mobilization

INTERVENTIONS:
Other: Exercise Movement Techniques based on mobilization — 10 sessions will be held twice a week, with each session taking an average of 50 minutes.
  Arms: Mobilization
Other: Exercise Movement Techniques based on stabilization — 10 sessions will be held twice a week, with each session taking an average of 50 minutes.
  Arms: Stabilization

SUMMARY:
Lumbar pain is one of the most common injuries being the cause of morbidity in the individual generating occupational disability with strong personal, social and economic impact. As one of the methods of treatment, Pilates is a method that has good results for the management of this dysfunction. However, it is not known exactly which approach Pilates can bring better results for this population. Therefore, the purpose of this study is to compare the effects of two types of Pilates method interventions on non-specific chronic low back pain.

A blinded randomized clinical trial, will be held. 28 patients divided randomly into two groups will be assessed, the Mobilization Pilates (MP) and the Stabilization Pilates (SP). Both groups will be formed by individuals of both sexes and aged 21 to 41 years with chronic low back pain. Both groups will receive 10 sessions of Pilates Methods twice a week, with each session taking an average of 50 minutes, therefore the MP will focus on a lumbo-pelvic mobilization exercises approach and the SP will focus on lumbo-pelvic stabilization exercises approach. At the beginning and end of the 5 weeks the individuals are evaluated to verify the presence of pain and disability with VAS of pain and Oswestry Questionnaire, and also with the Functional Movement Screen. Data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes aged between 21 and 40 years;
* Self-reported low back pain for at least 3 months;
* Disability Oswestry Index greater than 10%.

Exclusion Criteria:

* Diagnosis of pathognomonic low back pain caused by disc herniation with root involvement, inflammatory disorders, infections, osteoporosis, rheumatoid arthritis, fracture or tumor;
* Medical contraindication to the practice of Pilates;
* Childbirth or gestation in the last 6 months;
* Be performing any type of treatment for low back pain is medicated, physiotherapeutic or alternative during the period of intervention;
* Change the level of physical or sports activity during the intervention period;
* Participants who miss two sessions in a row or four sessions alternately without retrieving them in the same week will automatically be excluded from the survey; Or do not attend pre and post-test evaluation events.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-01-20 (Estimated)

PRIMARY OUTCOMES:
The change in Oswestry Low Back Disability Questionnaire | At the first session and 5 weeks after the intervention
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.
  The oswestry questionarie will be evaluated in the first session and after 5 weeks of Pilates training. So, the primary outcome is the change in the Oswestry score from baseline to 5 weeks.

SECONDARY OUTCOMES:
The change in Visual Analog Scale for Pain (VAS) | At the first session and 5 weeks after the intervention
  Pain intensity will be assessed using visual analog scale (VAS), which consists of a 10-cm horizontal line in which "0" means "No pain" and "10" means "The worst pain I can imagine". This visual analog scale for pain will be evaluated in the first session and after 5 weeks of Pilates training. So, this outcome is the change in VAS score from baseline to 5 weeks.
The change in The Functional Movement Screen (FMS) | At the first session and 5 weeks after the intervention
  The FMS is a screening for individuals who participate in physical activities by identifying limitations and restrictions in completing 7 movement tasks: deep squat, hurdle step, in-line lunch, shoulder mobility, active straight leg raise, trunk stability push-up, and rotatory stability.
  Each one of these 7 movement tasks are scored on a 0-3 ordinal scale. The FMS output is a single result given by summing each movement's score. The maximum score is 21. The lower the score, the higher is the patient's risk for injury.
  FMS will be evaluated before and after intervention. So, this outcome is the change in FMS score from baseline to 5 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson F Loss, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves de Araujo ME, Bezerra da Silva E, Bragade Mello D, Cader SA, Shiguemi Inoue Salgado A, Dantas EH. The effectiveness of the Pilates method: reducing the degree of non-structural scoliosis, and improving flexibility and pain in female college students. J Bodyw Mov Ther. 2012 Apr;16(2):191-8. doi: 10.1016/j.jbmt.2011.04.002. Epub 2012 Jan 5. PMID 22464116
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 1. N Am J Sports Phys Ther. 2006 May;1(2):62-72. PMID 21522216
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 2. N Am J Sports Phys Ther. 2006 Aug;1(3):132-9. PMID 21522225
- [Background] Cuchna JW, Hoch MC, Hoch JM. The interrater and intrarater reliability of the functional movement screen: A systematic review with meta-analysis. Phys Ther Sport. 2016 May;19:57-65. doi: 10.1016/j.ptsp.2015.12.002. Epub 2015 Dec 18. PMID 26777566
- [Background] Miyamoto GC, Costa LO, Cabral CM. Efficacy of the Pilates method for pain and disability in patients with chronic nonspecific low back pain: a systematic review with meta-analysis. Braz J Phys Ther. 2013 Nov-Dec;17(6):517-32. doi: 10.1590/S1413-35552012005000127. PMID 24346291
- [Background] Vigatto R, Alexandre NM, Correa Filho HR. Development of a Brazilian Portuguese version of the Oswestry Disability Index: cross-cultural adaptation, reliability, and validity. Spine (Phila Pa 1976). 2007 Feb 15;32(4):481-6. doi: 10.1097/01.brs.0000255075.11496.47. PMID 17304141